CLINICAL TRIAL: NCT02228135
Title: The Effect of Dexamethasone Dosing on Post-tonsillectomy Hemorrhage
Status: Completed | Type: Observational
Sponsor: Nicole Elsey (Other)
Responsible Party: Sponsor-Investigator, Nicole Elsey, Clinical Assistant Professor, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB14-00588
Record Dates: First submitted 2014-08-27; First posted 2014-08-28 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Tonsillectomy; Adenotonsillectomy
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non post-tonsillectomy hemorrhage: Children who do not have post-tonsillectomy hemorrhage.
  Interventions: Drug: Dexamethasone
- Post-tonsillectomy hemorrhage: Children return to the hospital after surgery with post-tonsillectomy hemorrhage.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone

SUMMARY:
This is a retrospective chart review looking at the effect of dexamethasone dosing on post-tonsillectomy hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a tonsillectomy
* Patients undergoing an adenotonsillectomy

Exclusion Criteria:

* All patients with a known history of bleeding or clotting disorders, as well as those patients who had presented to Nationwide Children's Hospital main operating room for control of PTH but had their initial tonsillectomy/adenotonsillectomy at an outlying facility will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children who have had tonsillectomy or adenotonsillectomy
Sampling Method: Non-Probability Sample
Enrollment: 9843 (Actual)
Dates: Start 2014-09; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Dexamethasone Dosage | once at start of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States